CLINICAL TRIAL: NCT06065930
Title: Mechanistic Studies in Human Subcutaneous Adipose Tissue
Brief Title: Adaptive Mechanisms In GRown up ObeSity Study (AMIGROS)
Acronym: AMIGROS
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02051-02
Record Dates: First submitted 2023-07-11; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Adipose cells; Fatty acids; Microdialysis; Stromal vascular fraction; Ectopic lipid accumulation; Fasting hyperinsulinemia; Insulin resistance; Amino acids
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, plasma, subcutaneous dialysates, urine, faeces and subcutaneous biopsy samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese insulin-sensitive subjects (Ob-IS): Obese Insulin Sensitive subjects (BMI > 30 kg/m2, fasting insulin < 9.0 mU/l and fasting plasma glucose < 6.1 mmol/l) undergoing subcutaneous microdialysis, needle biopsy, glucose clamp and MRI.
  Interventions: Device: Subcutaneous microdialysis
- Obese insulin-resistant subjects (Ob-IR): Obese Insulin Resistant subjects (BMI > 30 kg/m2, fasting insulin > 9.0 mU/l and fasting plasma glucose < 6.1 mmol/l) undergoing subcutaneous microdialysis, needle biopsy, glucose clamp and MRI.
  Interventions: Device: Subcutaneous microdialysis
- Lean healthy controls (Lean): Lean healthy controls (BMI < 25 kg/m2, fasting insulin < 9.0 mU/l and fasting plasma glucose < 6.1 mmol/l) undergoing subcutaneous microdialysis, needle biopsy, glucose clamp and MRI.
  Interventions: Device: Subcutaneous microdialysis

INTERVENTIONS:
Device: Subcutaneous microdialysis — Group with Ob-IS participants, collection of abdominal subcutaneous interstitial dialysates after an overnight´s fast for later measurements of metabolites and peptides eg galectin-1.
  Group with Ob-IR participants, collection of abdominal subcutaneous interstitial dialysates after an overnight´s fast for later measurements of metabolites and peptides eg galectin-1.
  Group with Leans, collection of abdominal subcutaneous interstitial dialysates after an overnight´s fast for later measurements of metabolites and peptides eg galectin-1.

SUMMARY:
The investigator recently showed that the glycan-binding adipokine galectin-1 increased during overfeeding and that galectin-1 independently could predict type 2 diabetes. Further, the molecules that induce insulin release in the fasting state when blood glucose is normal remain elusive. It is possible that galectin-1 is involved in adaptive mechanisms in adipose tissue in obese subjects.

DETAILED DESCRIPTION:
The investigator will define adaptive mechanisms in adipose tissue associated with galectin-1 in obese insulin-sensitive (Ob-IS) subjects compared with obese insulin-resistant (Ob-IR) subjects and lean healthy controls. Further, the investigator will study molecules secreted from adipose tissue that might trigger insulin secretion when blood glucose is normal.

The investigator hypothesizes that Ob-IS subjects keep fatty acid levels normal through an adaptive response in adipose tissue that involves up-regulation of galectin-1 for dampening of immune cell activity and stimulation of lipolysis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of age: 40.0 - 70.0 years
2. BMI: 18.0 - 25.0 kg/m2 (lean subjects) and BMI 30.0 - 38.0 kg/m2 (Ob-IS and Ob-IR)
3. Fasting insulin < 9.0 mU/l (lean and Ob-IS subjects) and fasting insulin > 9.0 mU/l (Ob-IR)
4. Fasting glucose < 6.1 mmol/l
5. Body temperature < 37.5°C
6. First-degree relative with known T2D in Ob-IR
7. Weight stable ± 5 kg < 3 months before screening
8. Fluent in Swedish and can follow given instructions
9. Consent given to participate

   Exclusion Criteria:
10. First-degree relative with known T2D in lean or Ob-IS subjects
11. Alcohol intake > 10 units/week or known high alcohol intake < 10 years back in time
12. Daily use of cigarettes or daily frequent use of smokeless tobacco not enabling the participant to suspend nicotine during a visit at the research center without getting abstinent
13. Regular physical activity corresponding to Saltin-Gimby level 4
14. Special diet eg Atkins or 5:2 for weight reduction. Vegetarian food accepted if duration > 1 year
15. Impaired fasting glucose (IFG) (venous fasting plasma glucose 6.1-6.9 mmol/l)
16. Type 2 diabetes according to ADA criteria
17. Ongoing or previous ischemic heart disease, eg angina pectoris, unstable angina or previous myocardial infarction treated with platelet inhibitors or non vitamin-K oral anticoagulants
18. Heart failure (NYHA II-IV) or cardiac arrhytmia that needs medical treatment
19. Previous cerebral infarction or transitory ischemic episodes (TIA) treated with platelet inhibitors or other anticoagulants
20. Peripheral arterial insufficiency eg claudication
21. Hypertension >170/105 mmHg at screening or more than one class of drugs for treatment of known hypertension
22. Lipid disorder defined as fasting serum triglycerides > 5.0 mmol/l or serum cholesterol > 7.5 mmol/l
23. Hematologic diseases such as anemia not being substituted (Hb < 130 g/l in males and Hv < 120 g/l in females) or disease causing bleeding disorder
24. Renal failure defined as absolute estimated glomerular filtration rate (eGFRcreatinine) < 60 ml/min/1.73 m2
25. Hypothyroidism defined as TSH > 4.0 mIE/l and symptoms
26. Liver disease e.g. hepatitis B, cirrhosis or conditions where AST or ALT are > 2 times UNL
27. Systemic inflammatory disease e.g. rheumatoid arthritis, ulcerative cholitis or Chrons disease. Celiac disease, dyspepsia or IBS are excepted
28. Chronic bronchitis or chronic obstructive pulmonary with disease symptoms
29. Previous pancreatitis or other disease in pancreas that needs treatment
30. Migraine elicited by stress
31. Spinal insufficiency causing inconvenience lying in supine position during the study day
32. Drug addiction interfering with the study procedures
33. Psychiatric insufficiency interfering with the study procedures
34. Medication with potential to affect adipose tissue metabolism that can not be stopped 10 days before the study days
35. Treatment with beta-blockers
36. Less than three months from previous use of antibiotics
37. Cancer disease < 5 years since diagnosis
38. Physical examination or laboratory results indicating that participation in the study is inappropriate
39. Pregnancy or intention to be pregnant during the study
40. Shift work > 1 time per week that might interfere with the circadian rhytm
41. Other reasons that causes the PI to believe that participation is inappropriate

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obese subjects and healthy lean controls will be recruited by advertisements in local newspapers and social media. Catchment area is western Sweden having about 1.5 million inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting galectin-1 concentration in subcutaneous interstitial fluid | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting Neuropilin-1 concentration in subcutaneous interstitial fluid | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment

SECONDARY OUTCOMES:
Fasting serum galectin-1 concentrations | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting serum neuropilin-1 concentrations | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting fatty acid levels in subcutaneous dialysates | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting plasma fatty acid concentrations | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting amino acid profile in subcutaneous dialysates | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Fasting serum amino acid concentrations | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Circulating metabolome including lipoprotein-related parameters measured by Mass Spectrometry | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Circulating lipidome including lipid derivatives measured by Mass Spectrometry | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Peptides identified by Mass Spectrometry in subcutaneous dialysates | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment
Ectopic lipid accumulation assessed by magnetic resonance imaging in relative measures | Nine weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 9 weeks after enrolment
RNA sequencing results of subcutaneous adipose cells | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Function of immune cells in subcutaneous stromal vascular fraction characterized by Fluorescence Activated Cell Sorting (FACS) | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Activation of insulin signaling proteins in adipose cells assessed by Western blot | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Function of microvascular endothelial cells in subcutaneous stromal vascular fraction | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Messenger RNA expression in whole adipose tissue | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Dysbiosis in faeces assessed by 16S rRNA gene sequencing | Six weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 6 weeks after enrolment
Metabolites in urine including acylcarnitines measured by Mass Spectrometry | Three weeks
  Comparison between eligible Ob-IS and Ob-IR subjects < 3 weeks after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders Jansson, Prof, Principal Investigator — Region Vastra Gotaland
Locations (1):
- Gothia Forum CTC, Gothenburg, Region Vastra Gotaland, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Sensitive personal data will be collected. Results will be shared if possible in the light of GDPR and other regulations, on an individual basis, after contact with the PI.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data analyses and completion of results for the major outcomes of the study will be 2025-2028. Data will be available for 15 years.
Access Criteria: Contact on an individual basis with PI of the study.

REFERENCES:
- [Result] Fryk E, Sundelin JP, Strindberg L, Pereira MJ, Federici M, Marx N, Nystrom FH, Schmelz M, Svensson PA, Eriksson JW, Boren J, Jansson PA. Microdialysis and proteomics of subcutaneous interstitial fluid reveals increased galectin-1 in type 2 diabetes patients. Metabolism. 2016 Jul;65(7):998-1006. doi: 10.1016/j.metabol.2016.04.003. Epub 2016 Apr 13. PMID 27282870
- [Result] Drake I, Fryk E, Strindberg L, Lundqvist A, Rosengren AH, Groop L, Ahlqvist E, Boren J, Orho-Melander M, Jansson PA. The role of circulating galectin-1 in type 2 diabetes and chronic kidney disease: evidence from cross-sectional, longitudinal and Mendelian randomisation analyses. Diabetologia. 2022 Jan;65(1):128-139. doi: 10.1007/s00125-021-05594-1. Epub 2021 Nov 7. PMID 34743218
- [Result] Fryk E, Olausson J, Mossberg K, Strindberg L, Schmelz M, Brogren H, Gan LM, Piazza S, Provenzani A, Becattini B, Lind L, Solinas G, Jansson PA. Hyperinsulinemia and insulin resistance in the obese may develop as part of a homeostatic response to elevated free fatty acids: A mechanistic case-control and a population-based cohort study. EBioMedicine. 2021 Mar;65:103264. doi: 10.1016/j.ebiom.2021.103264. Epub 2021 Mar 9. PMID 33712379
- [Result] Fryk E, Silva VRR, Jansson PA. Galectin-1 in Obesity and Type 2 Diabetes. Metabolites. 2022 Sep 30;12(10):930. doi: 10.3390/metabo12100930. PMID 36295832